CLINICAL TRIAL: NCT05100940
Title: Prospective Global Registry of Complications of Percutaneous Coronary Interventions
Brief Title: Progress Complication
Status: Recruiting | Type: Observational
Sponsor: Minneapolis Heart Institute Foundation (Other)
Responsible Party: Sponsor
Other Study IDs: PROGRESS-COMPLICATION
Record Dates: First submitted 2021-10-04; First posted 2021-10-29 (Actual); Last update posted 2021-10-29 (Actual); Status verified 2021-10

CONDITIONS: Coronary Artery Disease
Keywords: complications; Percutaneous Coronary intervention
MeSH Terms: conditions — Coronary Artery Disease | interventions — Cardiac Catheterization

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Cardiac Catheterization — Cardiac Catheterization

SUMMARY:
Coronary angiography and percutaneous coronary intervention (PCI) is often performed in patients with ischemic heart disease. The safety of PCI has improved with new devices and strategies, but complications still occur, especially during complex procedures. The objectives of this multi-center observational registry are to examine frequency of complications occuring during cardiac catheterization and PCI, examine procedural strategies utilized for complication management, and evaluate the clinical outcomes (both immediate and during follow-up.)

DETAILED DESCRIPTION:
The safety of PCI has improved with new devices and strategies, but complications still occur, especially during complex procedures. Systematic study of cardiac procedure complications can improve procedural safety and optimize short and long-term patient outcomes. The objectives of this multi-center observational registry are to

1-Examine the frequency and types of complications occurring during cardiac catheterization and PCI among participating sites, 2-Examine the procedural strategies (techniques and devices) utilized for complication management, 3-Evaluate the clinical outcomes (both immediate and during follow-up) after each complication type.

ELIGIBILITY:
* Over 18 years of age
* undergoing coronary angiography or PCI
* A complication occurred during or after the procedure

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Over 18 years of age and undergoing coronary angiography or PCI and a complication occurred during or after the procedure at each of the participating centers.
Sampling Method: Non-Probability Sample
Enrollment: 4000 (Estimated)
Dates: Start 2020-11-24 (Actual); Primary Completion 2030-12-31 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
in-hospital major cardiac adverse events (MACE) | From Date of Procedure to Date of Hospital Discharge, approximately 48-72 hrs after index procedure
  including any of the following adverse events prior to hospital discharge: death, stroke, myocardial infarction, recurrent angina requiring urgent repeat target vessel revascularization with PCI or coronary bypass surgery, and tamponade requiring pericardiocentesis or surgery.
Technical Success of PCI | From Date of Procedure to Date of Hospital Discharge, approximately 48-72 hrs after index procedure
  Technical success of PCI will be defined as successful lesion recanalization by any method with achievement of < 30% residual stenosis and TIMI 3 flow in both the main vessel and side branch. discharge: death, stroke, myocardial infarction, recurrent angina requiring urgent repeat target vessel revascularization with PCI or coronary bypass surgery, tamponade requiring pericardiocentesis or surgery); technical and procedural success; contrast volume, procedure time, fluoroscopy time, air kerma radiation dose.
Procedural success of PCI | From Date of Procedure to Date of Hospital Discharge, approximately 48-72 hrs after index procedure
  Procedural success of PCI will be defined as achievement of technical success and with no in-hospital major adverse cardiac events (MACE).

CONTACTS AND LOCATIONS:
Locations (1):
- Minneapolis Heart Institute Foundation, Minneapolis, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Mutlu D, Ser OS, Strepkos D, Carvalho PE, Alexandrou M, Kladou E, Mastrodemos O, Rangan BV, Sara JDS, Jalli S, Voudris K, Sandoval Y, Nicholas Burke M, Brilakis ES. Acute Kidney Injury Requiring Dialysis Following Percutaneous Coronary Intervention: Insights From the PROGRESS-COMPLICATIONS Registry. Catheter Cardiovasc Interv. 2025 Sep;106(3):1883-1891. doi: 10.1002/ccd.70012. Epub 2025 Jul 17. PMID 40676818